CLINICAL TRIAL: NCT02397109
Title: Study Of The Agreement Between The mDixon TSE Sequence And Conventional MRI Sequences In The Evaluation Of Dysimmune Orbitopathies
Brief Title: mDixon TSE MRI Sequence And Conventional MRI Sequences In Dysimmune Orbitopathies (DDX)
Acronym: DDX
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2015-1
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Dysthyroid Ophthalmopathies
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The dysthyroid orbitopathy (DO) is a chronic disease, evolving during 2 to 3 years, with a hypertrophy and a variable degree of inflammation of the eyelid muscles, the oculomotor muscles and the orbital fat.

If the diagnosis of OD is primarily clinical and laboratory, MRI is an additional contribution to the clinic, guiding the therapeutic management by detecting inflammatory lesions not found on clinical examination in 1/3 of cases.

The three MRI sequences conventionally practiced ((T2, T2-fat-sat, T1) allow muscles signal analysis oculomotor abnormalities as well as the orbital fat.

Compared to these sequences, the main advantage sequences DIXON is a faster acquisition. In addition, DIXON type of imaging overcomes most of these artifacts and to obtain a homogeneous fat removal.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 90 years, suffering from thyroid dysfunction proved by clinical and laboratory tests, with a bilateral clinical dysthyroid orbitopathy and undergoing an eye MRI

Exclusion Criteria:

* Absolute or relative contra-indication to MRI or to a contrast agent gadolinium injection (including pregnant or likely to be, breastfeeding women)
* Patient under guardianship
* Patient not willing to participate.
* Lack of affiliation to social security or medical state aid (AME) or universal health coverage (CMU)
* Motion artifact on the sequences, not corrected by the repeat sequences
* Metal artifact prohibiting the analysis of the region of interest

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a dysthyroid orbitopathy undergoing a MRI
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2015-04-04 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Assessment, by the determination of the Cohen's kappa coefficient, of the concordance between the conventional sequences (T1, T2, T2-fat-sat) and the mDIXON sequence for the diagnosis of inflammatory or non-inflammatory dysthyroid orbitopathy. | One hour

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France